CLINICAL TRIAL: NCT02924389
Title: Defining Antiretroviral Pharmacology Within HIV-1 Reservoirs of Males and Females
Brief Title: Dolutegravir in Reservoirs
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study terminated early due to the ongoing covid-19 pandemic making it unsafe to recruit participants for in-person visits. Participants are living with HIV who are antiretroviral therapy-naive and are at high risk of COVID-19 complications.
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cecile Delille Lahiri, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00089025; K23AI124913 (NIH)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: HIV
MeSH Terms: interventions — dolutegravir; abacavir, dolutegravir, and lamivudine drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anti-retroviral (ARV) Naïve Males (Other): Males diagnosed with HIV will undergo serial blood and tissue rectal sampling for twelve weeks after initiating ARV therapy as prescribed by their physician. Participants will be treated with either Triumeq or Truvada with dolutegravir.
  Interventions: Drug: dolutegravir; Drug: Triumeq; Drug: Truvada
- Anti-retroviral (ARV) Naïve Females (Other): Females diagnosed with HIV will undergo serial blood and tissue rectal sampling for twelve weeks after initiating ARV therapy as prescribed by their physician. Participants will be treated with either Triumeq or Truvada with dolutegravir.
  Interventions: Drug: dolutegravir; Drug: Triumeq; Drug: Truvada

INTERVENTIONS:
Drug: dolutegravir — Tivicay is a human immunodeficiency virus type 1 (HIV-1) integrase strand transfer inhibitor (INSTI) indicated in combination with other antiretroviral agents for the treatment of HIV-1 infection. 50 mg of Tivicay (dolutegravir) will be taken orally once a day.
  Other Names: Tivicay
Drug: Triumeq — Triumeq is a fixed-dose combination drug for the treatment of HIV/AIDS. It is a combination of 600 mg abacavir, 50 mg dolutegravir and 300 mg lamivudine. Triumeq will be taken orally once daily.
Drug: Truvada — Truvada is a combination of emtriva and viread, both nucleoside analog HIV-1 reverse transcriptase inhibitors. Truvada is indicated in combination with other antiretroviral agents for the treatment of HIV-1 infection. One Truvada tablet (containing 200 mg/300 mg of emtricitabine and tenofovir disoproxil fumarate) will be taken orally once daily.

SUMMARY:
The purpose of this study is to find out how well the HIV medication dolutegravir gets into different parts of the body including blood plasma, special blood cells, and rectal tissue. Specifically, investigators want to compare how fast dolutegravir lowers the HIV viral load in these three different sites. In addition, as an exploratory aim, investigators seek to learn if there are any differences in how dolutegravir acts in males and females. Results of this study will provide more information about HIV medications and their limitations. In the future, this could help create better HIV medications that can get into these hard-to-reach places and eventually cure HIV infection.

DETAILED DESCRIPTION:
Emerging evidence indicates that sites outside of blood plasma, such as peripheral blood mononuclear cells (PBMCs) and gut-associated lymphoid tissue, remain reservoirs for HIV and play critical roles in viral persistence despite long-term potent combination antiretroviral therapy (cART). Suboptimal ARV drug concentrations within these reservoirs are thought to contribute to our inability to fully eradicate HIV. In addition, host factors such as sex have been found to impact ARV drug exposure within these sites and effect key outcomes such as time to virologic suppression. The understanding of reservoir site pharmacology and the impact on sex is limited due to several barriers: 1) Difficulty in sampling reservoir sites intensively and 2) Scarcity of women enrolled in HIV clinical research studies. Optimal drug concentrations are ideally determined early in drug development by dose-ranging studies that require intensive blood plasma sampling; this methodology is impractical to employ within tissue sites. To mitigate these barriers, the researchers propose to study the pharmacology of the integrase strand transfer inhibitor dolutegravir (DTG) within three body compartments: blood plasma, PBMCs, and rectal tissue using a novel integrated population pharmacokinetic-viral dynamic (PK-VD) modeling approach. This PK-VD modeling strategy generates concentration-response relationships with limited sampling and dosing simulations ideally suited to reservoir sites.

The primary aim of this study is to validate the integrated population PK-VD model that quantitatively describes the relationship between dolutegravir (DTG) exposure and HIV viral decay in blood plasma. The second aim of this study is to develop an integrated population pharmacokinetic-viral dynamic (PK-VD) model to describe the relationship between DTG exposure and HIV viral decay in peripheral blood mononuclear cells and rectal tissue reservoir sites. The third aim is exploratory and will investigate sex differences in DTG penetration into blood plasma, peripheral blood mononuclear cells and rectal tissue reservoirs reservoirs as well as its impact on the rectal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* No ARVs in the last 6 months (from date of screening)
* No documented or suspected resistance to integrase inhibitors (dolutegravir, elvitegravir, raltegravir, or bictegravir).
* Creatinine Clearance >50 mL/min, as calculated by the Cockcroft-Gault equation within 90 days of screen
* Liver function testing, including alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase < 5 times upper limit of normal within 90 days of screen
* Intact gastrointestinal tract
* Able and willing to give informed consent
* Willing and eligible to initiate ARV therapy with Triumeq, DTG + Truvada (TDF/FTC), or DTG + Descovy (FTC/TAF)
* Agree to receive from their provider and pay for a prescribed supply of the drug, Tivicay® (dolutegravir/DTG), with either Triumeq, or Truvada or Descovy as determined by their primary HIV provider

  * Agree to take the prescribed medication by mouth
  * Agree that they (the participant) is responsible for bringing these medications with them to their study visits
* Willing to undergo serial blood and rectal tissue sampling
* Female participants' must be willing to have a pregnancy test done at each visit. Female participants of childbearing potential (FCB) must agree to either commit to continued abstinence from heterosexual intercourse or to use a reliable form of birth control such as oral contraceptive pills, intrauterine device, Nexplanon, DepoProvera, permanent sterilization, or another acceptable method, as determined by the investigator for the duration of the study. FCB are defined as sexually mature women who have not undergone hysterectomy or bilateral oophorectomy or have not been naturally postmenopausal for at least 24 consecutive months (i.e have had menses at any time in preceding 24 months)

Exclusion Criteria:

* Pregnant or attempting to conceive now or during the course of the study
* Self-reported or documented current anal or rectal disease prohibiting safe anoscopy and biopsies, in investigator's opinion.
* Taking concurrent medications that interfere with DTG
* Bleeding diathesis
* Platelet count <50,000 mm3
* Medical condition that interferes with conduct of study, in investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Lahiri, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Health System, Atlanta, Georgia
  - Ponce De Leon Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lahiri CD, Brown NL, Ryan KJ, Acosta EP, Sheth AN, Mehta CC, Ingersoll J, Ofotokun I. HIV RNA persists in rectal tissue despite rapid plasma virologic suppression with dolutegravir-based therapy. AIDS. 2018 Sep 24;32(15):2151-2159. doi: 10.1097/QAD.0000000000001945. PMID 30005011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began September 2016 and all follow up was complete by September 11, 2019. Participants were enrolled at the Grady Ponce de Leon Center and Grady Health System in Atlanta, Georgia, USA.
Groups:
- Anti-retroviral (ARV) Naïve Males: Males diagnosed with HIV undergoing serial blood and tissue rectal sampling for twelve weeks after initiating anti-retroviral (ARV) therapy as prescribed by their physician. Participants were treated with either Triumeq (abacavir 600 mg/dolutegravir 50 mg/lamivudine 300 mg), or Truvada (emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg) plus and dolutegravir (50 mg), or Descovy (emtricitabine 200 mg/tenofovir alafenamide 25 mg) plus dolutegravir (50 mg).
- Anti-retroviral (ARV) Naïve Females: Females diagnosed with HIV undergoing serial blood and tissue rectal sampling for twelve weeks after initiating ARV therapy as prescribed by their physician. Participants were treated with either Triumeq (abacavir 600 mg/dolutegravir 50 mg/lamivudine 300 mg), or Truvada (emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg) plus and dolutegravir (50 mg), or Descovy (emtricitabine 200 mg/tenofovir alafenamide 25 mg) plus dolutegravir (50 mg).
Period: Overall Study
Arm/Group | Anti-retroviral (ARV) Naïve Males | Anti-retroviral (ARV) Naïve Females
Started | 16 | 6
Completed | 8 | 6
Not Completed | 8 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Participant began ARVs prior to study intervention | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Anti-retroviral (ARV) Naïve Males: Males diagnosed with HIV undergoing serial blood and tissue rectal sampling for twelve weeks after initiating ARV therapy as prescribed by their physician. Participants were treated with either Triumeq (abacavir 600 mg/dolutegravir 50 mg/lamivudine 300 mg), or Truvada (emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg) plus and dolutegravir (50 mg), or Descovy (emtricitabine 200 mg/tenofovir alafenamide 25 mg) plus dolutegravir (50 mg).
- Total: Total of all reporting groups
Arm/Group | Anti-retroviral (ARV) Naïve Males | Anti-retroviral (ARV) Naïve Females | Total
Number analyzed (Participants) | 16 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (9.8) | 45.6 (8.0) | 38.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 16 | 0 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 5 | 19
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Dolutegravir Concentration
Description: Dolutegravir concentrations in blood plasma are assessed as the maximum dolutegravir concentration (Cmax) and 24 hour trough (lowest) concentration (C24h) of dolutegravir in micrograms per milliliter (µg/mL). Blood samples for pharmacokinetics were obtained prior to dosing (hour 0) and 1, 2, 3, 4, 6, 8, and 24 hours after dosing.
Time Frame: Day 84 (hour 0 through 24)
Population: This analysis includes participants who completed at least one study visit. Fourteen participants completed all study visits and 2 completed a portion of study visits. Males and females are combined for all primary and secondary analyses and are separated only for exploratory study outcomes.
Measure: Median (Inter-Quartile Range); unit: µg/mL
Groups:
- Anti-retroviral (ARV) Naïve Males and Females: Males and females diagnosed with HIV undergoing serial blood and tissue rectal sampling for twelve weeks after initiating ARV therapy as prescribed by their physician. Participants were treated with either Triumeq (abacavir 600 mg/dolutegravir 50 mg/lamivudine 300 mg), or Truvada (emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg) plus and dolutegravir (50 mg), or Descovy (emtricitabine 200 mg/tenofovir alafenamide 25 mg) plus dolutegravir (50 mg).
Arm/Group | Anti-retroviral (ARV) Naïve Males and Females
Number analyzed (Participants) | 16
µg/mL
  First-dose pharmacokinetics (Cmax) | 2.01 [1.17 to 2.32]
  Steady state pharmacokinetics (Cmax) | 2.34 [1.84 to 3.04]
  Trough dolutegravir concentration (C24h) | 0.56 [0.44 to 1.21]

2. Secondary Outcome: Dolutegravir Exposure in Peripheral Blood Mononuclear Cells (PBMC)
Description: Dolutegravir concentrations in peripheral blood mononuclear cells required for HIV viral load decline.
Time Frame: Up to Day 84
Population: Due to lack of viral dynamic decline in PBMCs and inability to measure intracellular dolutegravir consistently with the assays, this secondary outcome could not be assessed.
Arm/Group | Anti-retroviral (ARV) Naïve Males and Females
Number analyzed (Participants) | 0

3. Secondary Outcome: Dolutegravir Concentration in Rectal Tissue
Description: Rectal dolutegravir concentrations in rectal tissue stratified by virologic suppressors vs non-suppressors.
Time Frame: Week 2, Week 6, Week 12
Population: This analysis includes the first 12 study participants; the analysis was not extended to subsequent participants due to study findings being sufficient from the first 12 participants. One participant was removed from this analysis because they had undetectable virus in rectal tissue at the baseline assessment.
Measure: Median (Full Range); unit: ng/mL
Groups:
- HIV RNA Suppressors: Males and females diagnosed with HIV undergoing serial blood and tissue rectal sampling for twelve weeks after initiating ARV therapy as prescribed by their physician. Suppressors are participants with baseline detectable rectal tissue HIV RNA who achieved rectal tissue HIV RNA suppression at any time point during the 12 week study.
- HIV RNA Non-suppressors: Males and females diagnosed with HIV undergoing serial blood and tissue rectal sampling for twelve weeks after initiating ARV therapy as prescribed by their physician. Non-suppressors are participants with baseline detectable rectal tissue HIV RNA who did not achieve rectal tissue HIV RNA suppression during the 12 week study.
Arm/Group | HIV RNA Suppressors | HIV RNA Non-suppressors
Number analyzed (Participants) | 3 | 8
ng/mL
  Week 2 | 1606 [1420 to 1791] | 749 [608 to 1559]
  Week 6 | 724 [102 to 1579] | 625 [134 to 1452]
  Week 12 | 473 [163 to 12369] | 373 [2.65 to 621]

4. Primary Outcome: Time of Maximum Dolutegravir Concentration
Description: Time of maximum dolutegravir concentration is assessed in hours for the time periods of after the first dose and during steady state. Blood samples for pharmacokinetics were obtained prior to dosing (hour 0) and 1, 2, 3, 4, 6, 8, and 24 hours after dosing.
Time Frame: Day 84 (hour 0 through 24)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Anti-retroviral (ARV) Naïve Males and Females
Number analyzed (Participants) | 16
hours
  First-dose pharmacokinetics (Tmax) | 1.5 [1.0 to 3.8]
  Steady state pharmacokinetics (Tmax) | 3.0 [3.0 to 4.0]

5. Primary Outcome: Area Under the Dolutegravir Plasma Concentration vs Time Curve
Description: The area under the dolutegravir plasma concentration vs time curve in a 24 hour period (AUC24h) is assessed in hours times micrograms per millimeters (h* µg/mL) for the time periods of after the first dose and during steady state. Blood samples for pharmacokinetics were obtained prior to dosing (hour 0) and 1, 2, 3, 4, 6, 8, and 24 hours after dosing.
Time Frame: Day 84 (hour 0 through 24)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: h* µg/mL
Arm/Group | Anti-retroviral (ARV) Naïve Males and Females
Number analyzed (Participants) | 16
h* µg/mL
  First-dose pharmacokinetics (AUC24h) | 22.30 [15.03 to 30.85]
  Steady state pharmacokinetics (AUC24h) | 27.24 [24.48 to 48.08]

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time consent was given to participate in the study through the final study visit at Day 84.
Arm/Group | Anti-retroviral (ARV) Naïve Males | Anti-retroviral (ARV) Naïve Females
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6
Other Adverse Events (participants affected / at risk) | 9/16 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-retroviral (ARV) Naïve Males (N=16) | Anti-retroviral (ARV) Naïve Females (N=6)
Rectal bleeding (Surgical and medical procedures) | 5 | 3
Rectal/anal pain (Surgical and medical procedures) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Fatigue (General disorders) | 0 | 2
Nausea (General disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Night sweats (General disorders) | 1 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 1
Lymphadenopathy (Infections and infestations) | 1 | 2
Weight gain (General disorders) | 0 | 1
Genital herpes simplex (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Oral ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT02924389/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT02924389/ICF_000.pdf